CLINICAL TRIAL: NCT02116361
Title: BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex as Treatment for Major Depressive Disorder in Adult Females
Brief Title: OnabotulinumtoxinA as Treatment for Major Depressive Disorder in Adult Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-135
Record Dates: First submitted 2014-04-15; First posted 2014-04-16 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo for onabotulinumtoxinA 50 U (Placebo Comparator): Placebo (normal saline) for onabotulinumtoxinA 50 U injected into protocol-specified areas on Day 1.
  Interventions: Drug: Normal Saline
- onabotulinumtoxinA 50 U (Experimental): OnabotulinumtoxinA 50 U injected into protocol-specified areas on Day 1.
  Interventions: Biological: onabotulinumtoxinA
- Placebo for onabotulinumtoxinA 30 U (Placebo Comparator): Placebo (normal saline) for onabotulinumtoxinA 30 U injected into protocol-specified areas on Day 1.
  Interventions: Drug: Normal Saline
- onabotulinumtoxinA 30 U (Experimental): OnabotulinumtoxinA 30 U injected into protocol-specified areas on Day 1.
  Interventions: Biological: onabotulinumtoxinA

INTERVENTIONS:
Biological: onabotulinumtoxinA — OnabotulinumtoxinA injected into protocol-specified areas on Day 1.
  Other Names: BOTOX®; botulinum toxin Type A
  Arms: onabotulinumtoxinA 30 U; onabotulinumtoxinA 50 U
Drug: Normal Saline — Placebo (normal saline) injected into protocol-specified areas on Day 1.
  Arms: Placebo for onabotulinumtoxinA 30 U; Placebo for onabotulinumtoxinA 50 U

SUMMARY:
This study will evaluate the safety and efficacy of onabotulinumtoxinA (BOTOX®) compared with placebo as treatment for major depressive disorder (MDD) in adult females.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe major depressive disorder

Exclusion Criteria:

* Prior treatment with botulinum toxin of any serotype for any reason
* Use of antidepressant medication for depression within 2 weeks of study
* Diagnosis of Myasthenia gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2014-04-22 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shobhal Patel, Study Director — Allergan
Locations (35):
- United States (35):
  - Woodland International Research Group, Little Rock, Alaska
  - CITrials, Bellflower, California
  - Radiant Research/Comprehensive Clinical Development, Inc., Cerritos, California
  - Collaborative Neuroscience Network Inc., Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Excell Research, Inc., Oceanside, California
  - NRC Research Institute, Orange, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Compass Research LLC-North Clinic, Leesburg, Florida
  - Research Centers of America, LLC, Oakland Park, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Uptown Research Institute, LLC, Chicago, Illinois
  - Psychiatric Medicine Associates, LLC, Skokie, Illinois
  - St. Louis Clinical Trials, LLC, St Louis, Missouri
  - Integrative Clinical Trials, Brooklyn, New York
  - SPRI Clinical Trials, Brooklyn, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Clinical Neuroscience Solutions, INC, Memphis, Tennessee
  - KRK Medical Research, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Virginia Commonwealth University Clinical Research Services Unit, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Zain Research LLC, Richland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brin MF, Durgam S, Lum A, James L, Liu J, Thase ME, Szegedi A. OnabotulinumtoxinA for the treatment of major depressive disorder: a phase 2 randomized, double-blind, placebo-controlled trial in adult females. Int Clin Psychopharmacol. 2020 Jan;35(1):19-28. doi: 10.1097/YIC.0000000000000290. PMID 31609787

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Normal Saline) for onabotulinumtoxinA 50 U: Placebo (normal saline) for onabotulinumtoxinA 50 U injected into protocol-specified areas on Day 1.
- Placebo (Normal Saline) for onabotulinumtoxinA 30 U: Placebo (normal saline) for onabotulinumtoxinA 30 U injected into protocol-specified areas on Day 1.
Period: Overall Study
Arm/Group | Placebo (Normal Saline) for onabotulinumtoxinA 50 U | onabotulinumtoxinA 50 U | Placebo (Normal Saline) for onabotulinumtoxinA 30 U | onabotulinumtoxinA 30 U
Started | 69 | 65 | 59 | 65
Completed | 38 | 34 | 33 | 34
Not Completed | 31 | 31 | 26 | 31
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 2
Not completed — Physician Decision | 2 | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 3
Not completed — Other Reasons | 3 | 3 | 3 | 3
Not completed — Lack of Efficacy | 5 | 7 | 4 | 3
Not completed — Lost to Follow-up | 4 | 5 | 7 | 5
Not completed — Personal Reasons | 6 | 6 | 4 | 9
Not completed — Investigator Decision - Relapse | 9 | 7 | 8 | 5

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat: Enrolled subjects who received treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Normal Saline) for onabotulinumtoxinA 50 U | onabotulinumtoxinA 50 U | Placebo (Normal Saline) for onabotulinumtoxinA 30 U | onabotulinumtoxinA 30 U | Total
Number analyzed (Participants) | 67 | 65 | 58 | 65 | 255
Age, Customized [Number; unit: Participants]
  <40 years | 26 | 21 | 21 | 26 | 94
  ≥ 40 years | 41 | 44 | 37 | 39 | 161
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 65 | 58 | 65 | 255
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Baseline Values for the Clinic 10-Item Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item scale completed by clinic personnel that assesses the subject's symptoms of depression. Each question is answered on a 7-point scale ranging from no symptoms to worst possible symptoms. The total score is summed for all responses and ranges from 0 to 60. A negative change from baseline indicates an improvement in symptoms and a positive change from baseline indicates a worsening.
Time Frame: Baseline
Population: Modified Intent to Treat: Enrolled subjects who received treatment with data at the noted time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Normal Saline) for onabotulinumtoxinA 30 U | onabotulinumtoxinA 30 U | Placebo (Normal Saline) for onabotulinumtoxinA 50 U | onabotulinumtoxinA 50 U
Number analyzed (Participants) | 58 | 65 | 67 | 65
Scores on a Scale | 31.4 (3.99) | 32.0 (4.12) | 32.4 (5.34) | 32.0 (4.44)

2. Primary Outcome: Change From Baseline Values in the Clinic 10-Item Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: as for outcome 1
Time Frame: Week 6
Population: Modified Intent to Treat: Enrolled subjects who received treatment with data at the noted time point
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo (Normal Saline) for onabotulinumtoxinA 30 U | onabotulinumtoxinA 30 U | Placebo (Normal Saline) for onabotulinumtoxinA 50 U | onabotulinumtoxinA 50 U
Number analyzed (Participants) | 58 | 65 | 67 | 65
Scores on a Scale | -7.9 (1.4) | -11.6 (1.4) | -12.9 (1.2) | -11.5 (1.2)

3. Secondary Outcome: Baseline Values for the 7-Item Clinical Global Impression of Severity of Illness (CGI-S) Score
Description: The CGI-S is a 7-point scale assessed by the clinician to rate the severity of the subject's symptoms. Scores range from 1 to 7, from normal (1, not at all ill) to among the most extremely ill patients (7). A negative change from baseline indicates an improvement in symptoms and a positive change from baseline indicates a worsening.
Time Frame: Baseline
Population: Modified Intent to Treat: Enrolled subjects who received treatment with data at the noted time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Normal Saline) for onabotulinumtoxinA 30 U | onabotulinumtoxinA 30 U | Placebo (Normal Saline) for onabotulinumtoxinA 50 U | onabotulinumtoxinA 50 U
Number analyzed (Participants) | 58 | 65 | 67 | 65
Scores on a Scale | 4.2 (0.43) | 4.4 (0.53) | 4.4 (0.53) | 4.5 (0.50)

4. Secondary Outcome: Change From Baseline Values in the 7-Item Clinical Global Impression of Severity of Illness (CGI-S) Score
Description: as for outcome 3
Time Frame: 24 Weeks
Population: Modified Intent to Treat: Enrolled subjects who received treatment with data at the noted time point
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo (Normal Saline) for onabotulinumtoxinA 30 U | onabotulinumtoxinA 30 U | Placebo (Normal Saline) for onabotulinumtoxinA 50 U | onabotulinumtoxinA 50 U
Number analyzed (Participants) | 33 | 36 | 38 | 34
Scores on a Scale | -1.4 (0.2) | -1.9 (0.2) | -2.6 (0.2) | -2.9 (0.2)

5. Secondary Outcome: Baseline Values in the Clinic Hamilton Depression Rating Scale 17-Item Version (HAM-D17)
Description: The HAM-D17 is assessed by the clinician based on subject interview. The total scores range from 0 to 53. A higher total score indicates more severe depression. A negative change from baseline indicates an improvement in symptoms and a positive change from baseline indicates a worsening.
Time Frame: Baseline
Population: Modified Intent to Treat: Enrolled subjects who received treatment with data at the noted time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Normal Saline) for onabotulinumtoxinA 30 U | onabotulinumtoxinA 30 U | Placebo (Normal Saline) for onabotulinumtoxinA 50 U | onabotulinumtoxinA 50 U
Number analyzed (Participants) | 58 | 65 | 67 | 65
Scores on a Scale | 23.7 (3.15) | 24.5 (3.03) | 23.3 (2.94) | 23.0 (3.32)

6. Secondary Outcome: Change From Baseline Values in the Clinic Hamilton Depression Rating Scale 17-Item Version (HAM-D17)
Description: as for outcome 5
Time Frame: 24 Weeks
Population: Modified Intent to Treat: Enrolled subjects who received treatment with data at the noted time point
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo (Normal Saline) for onabotulinumtoxinA 30 U | onabotulinumtoxinA 30 U | Placebo (Normal Saline) for onabotulinumtoxinA 50 U | onabotulinumtoxinA 50 U
Number analyzed (Participants) | 33 | 36 | 38 | 34
Scores on a Scale | -11.5 (1.1) | -13.4 (1.1) | -16.1 (0.8) | -17.4 (0.8)

ADVERSE EVENTS:
Description: The Safety Population was used to assess AEs and SAEs and consisted of all randomized patients who received at least 1 injection of the study treatment
Arm/Group | Placebo (Normal Saline) for onabotulinumtoxinA 50 U | onabotulinumtoxinA 50 U | Placebo (Normal Saline) for onabotulinumtoxinA 30 U | onabotulinumtoxinA 30 U
Serious Adverse Events (participants affected / at risk) | 5/67 | 0/65 | 1/58 | 3/65
Other Adverse Events (participants affected / at risk) | 21/67 | 18/65 | 10/58 | 21/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Normal Saline) for onabotulinumtoxinA 50 U (N=67) | onabotulinumtoxinA 50 U (N=65) | Placebo (Normal Saline) for onabotulinumtoxinA 30 U (N=58) | onabotulinumtoxinA 30 U (N=65)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hallucination, Auditory (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 1
Varicose Vein (Vascular disorders) | 1 | 0 | 0 | 0
Sudden Death (General disorders) | 0 | 0 | 0 | 1
Benign Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Normal Saline) for onabotulinumtoxinA 50 U (N=67) | onabotulinumtoxinA 50 U (N=65) | Placebo (Normal Saline) for onabotulinumtoxinA 30 U (N=58) | onabotulinumtoxinA 30 U (N=65)
Sinusitis (Infections and infestations) | 0 | 0 | 4 | 4
URI (Infections and infestations) | 3 | 4 | 1 | 3
Headache (Nervous system disorders) | 15 | 11 | 4 | 9
Eyelid Ptosis (Eye disorders) | 0 | 2 | 0 | 4
Nasopharyngitis (Infections and infestations) | 6 | 3 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.